CLINICAL TRIAL: NCT05719987
Title: Effect of Biodentine Application as an Apical Plug on the Healing of Apical Lesions on Immature Permanent Molars.
Brief Title: Biodentine as an Apical Plug in Immature Permanent Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UDDS-Pedo-12-2016
Record Dates: First submitted 2022-02-10; First posted 2023-02-09 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Periapical Periodontitis
Keywords: Apexification; MTA; Biodentine; Immature molars
MeSH Terms: conditions — Periapical Periodontitis | interventions — tricalcium silicate; Pemetrexed

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple Masking: Patients, Investigators and Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biodentine Group (Experimental): study group
  Interventions: Other: Biodentine
- MTA Group (Other): control group
  Interventions: Other: MTA

INTERVENTIONS:
Other: Biodentine — After the endodontic procedure, Biodentine will be placed into the apical portion of the canals. After 12 min, the coronal and middle third of the root canal will be filled with gutta-percha and AH Plus. The coronal restoration will be completed with GIC, composite, and stainless-steel crown.
  Arms: Biodentine Group
Other: MTA — After the endodontic procedure, MTA will be placed into the apical portion of the canals. After 12 min, the coronal and middle third of the root canal will be filled with gutta-percha and AH Plus. The coronal restoration will be completed with GIC, composite, and stainless-steel crown.
  Arms: MTA Group

SUMMARY:
Following the randomization procedure, patients will be divided into 2 groups (12 immature molars in each group): Group I will be treated with MTA as apical plug, whereas group II will be treated with Biodentine as apical plug. After working length determination, instrumentation and sterilizing root canals, apical plug will be done as following:

Biodentine Group: Biodentine will be placed into the apical portion of canals. After 12 min the coronal and middle third of the root canal will be filled with gutta-percha and AH Plus. The coronal restoration will be completed with GIC, composite, and stainless-steel crown.

MTA Group: MTA will be placed into the apical portion of canals, then a moist cotton pellet will be placed and the access cavity will be restored with temporary filling. Next day, temporary filling and the cotton pellet will be removed, then the coronal restoration will be performed as Biodentine group.

Patients of both groups will be recalled for clinical and radiographical follow-up within 12 months after treatment.

DETAILED DESCRIPTION:
Following the randomization procedure, patients will be assigned sequential numbers in the order of enrolment. Group I will include 12 immature molars treated with MTA (White ProRoot MTA, Dentsply, Tulsa, OK, USA) as apical plug, whereas group II will include 12 immature molars treated with Biodentine (Septodont, Saint-Maur-des-Fosses, France) as apical plug. All the apexification treatments will be performed by the researcher. Under local anesthesia and rubber dam isolation, all superficial caries will be removed with carbide fissure bur mounted on a low-speed hand-piece. Access cavity will be prepared using an endo-z bur mounted on high-speed hand-piece, and the cavity will be rinsed with 2.5% NaOCl. Working length will be calculated radiographically with K-files (Mani, INK, Japan) and recorded as reference. root canals will be instrumented gently with Fanta AF3 (Fanta Dental Materials Co., LTD, Shanghai, China) and copious irrigation with 1.3% sodium hypochlorite (NaOCI) (Merck, Darmstadt, Germany) by a 30- gauge endodontic irrigating needle (Sybron Endo, Crop, Orange, CA, USA). As final irrigation all canals will be filled up with NaOCl 1.3% and activated with #40 U-file ultrasonic tip (Zipperer Co., Munchen, Germany) for 30 seconds for each canal, then all canals will be irrigated with normal saline, then all canals will be filled up with Q-mix (Dentsply Tulsa Dental, Tulsa, OK, USA) and activated with #40 U-file ultrasonic tip (Zipperer Co., Munchen, Germany) for 10 seconds. After drying with large sterile paper points apical plug will be done according to randomization MTA with 2 visits or Biodentine with one visit.

Biodentine Group (performed in a single clinic visit of approximately 45 minutes): Biodentine will be placed with MAP-One System (Produits Dentaires, sa vevey, switzerland) into the apical portion of canals with about 4 mm thickness and adapted to the canal walls with an endodontic hand plugger (Dentsply, Tulsa, OK, USA). Correct placement of the Biodentine plugs will be verified with a radiograph. After 12 min the setting of Biodentine will be detected gently with #40 k-file (Mani, INK, Japan). The coronal and middle third of the root canal will be filled with gutta-percha in conjunction with AH Plus sealer (Dentsply Sirona Endodontics) using lateral condensation technique. The coronal restoration will be completed with GIC Fuji IX (GC Corporation, Tokyo, Jappan), then bonded resin composite (3M ESPE, Dental Products, St. Paul, MN, USA), and stainless-steel crown (3M ESPE, Dental Products, St. Paul, MN, USA).

MTA Group (performed in 2 clinic visits, each visit will be approximately 30 minutes): MTA will be placed with MAP-One System (Produits Dentaires, sa vevey, switzerland) into the apical portion of canals with about 4 mm thickness and adapted to the canal walls with an endodontic hand plugger (Dentsply, Tulsa, OK, USA). Correct placement of the MTA plugs will be verified with a radiograph. After inserting MTA, a moist cotton pellet will be placed in the canal, and the access cavity will be restored with temporary filling (TG, Germany). Next day, under local anesthesia and rubber dam isolation, the temporary filling and the cotton pellet will be removed and the setting of MTA will be detected gently with #40 k-file (Mani, INK, Japan). The coronal and middle third of the root canal will be filled with gutta-percha in conjunction with AH Plus sealer (Dentsply Sirona Endodontics) using lateral condensation technique. The coronal restoration will be completed with GIC Fuji IX (GC Corporation, Tokyo, Jappan), then bonded resin composite (3M ESPE, Dental Products, St. Paul, MN, USA), and stainless steel crown (3M ESPE, Dental Products, St. Paul, MN, USA).

Patients of both groups will be recalled for radiographical follow-up after the end of treatment at 1, 3, 6 and 12 months. Periapical radiographs will be obtained under standard exposure conditions (60 kVp, 7 mA and 0.32 s) using a dental X-ray machine (Gendex GX, Lake Zurich, IL, USA) and intraoral sensor (VATECH. Gyeonggi-do, Korea) . The radiographic assessment will be done with two pre-trained independent investigators. Each investigator will determine the size of apical lesion using "Image J" program and scored in both groups blindly, independently and will repeat the radiographic scoring after 1 month to assess the intraobserver reliability. Any disagreement on apical lesion size for a particular root resulted in joint evaluation until agreement will be reached.

Patients of both groups will be recalled for clinical follow-up after the end of treatment at 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months, 12 months to detect pain, swelling, tenderness to percussion, abscess, fistula, and abnormal tooth mobility Finally, the numerical data of the apical lesions sizes and ranked data of clinical variables will be statistically analyzed using SPSS, and any statistically significant values will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children.
* Healthy children without any systemic disease or compromised immune status.
* Children with first immature mandibular molar with at least one canal sized #60 or more with an apical lesion.

Exclusion Criteria:

* Patients with advanced periodontitis (more than 5 mm periodontal attachment and bone loss).
* Molars that cannot be restored (root fracture, unrestorable tooth, massive internal or external).
* Molars that had previous endodontic treatment.

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the apical lesion size | after 1,3,6 and 12 months of root canal obturation
  The apexification procedure was judged to be radiographically successful if it demonstrated the following criteria: (1) reduction of apical lesion size (2) Normal periodontal ligament space (2) No furcation pathosis, and (3) No external resorption.
  The apexification procedure was judged to be radiographically unsuccessful if the apical lesion size increased.
  The apexification procedure was judged to be doubtful if the apical lesion size didn't change
Change in the clinical assessment of success | 1 day, 3 days, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months of root canal obturation
  The apexification procedure was decided a clinical success if the tooth fulfilled the following criteria: (1) No pain, (2) No swelling, (3) No tenderness to percussion, (4) No abscess or fistula, and (5) No abnormal tooth mobility.

SECONDARY OUTCOMES:
Change in the apical lesion healing speed | after 1,3,6 and 12 months of root canal obturation
  Apical lesion healing speed of MTA apical plugs and Biodentine apical plugs in necrotic immature permanent molars with apical lesions using "Image J" to determine the percentage of apical lesion reduction
Change in the periapical index (PAI) | after 1,3,6 and 12 months of root canal obturation
  Radio-graphically, the periapical index provides an ordinal scale of 5 scores ranging from ''healthy'' to ''severe periodontitis with exacerbating features''. (1) Normal periapical structures. (2) Small changes in bone structure. (3) Changes in bone structure with some diffuse mineral loss. (4) Periodontitis with well-deﬁned radiolucent area. (5) Severe periodontitis with exacerbating features. (1, 2: healthy and 3, 4, 5: pathological).

CONTACTS AND LOCATIONS:
Overall Officials: Chaza Kouchaji, Professor, Study Director — supervisal; Thuraya Lazkani, Professor, Study Director — co-supervisal
Locations (1):
- College of dentistry., Damascus, Al-Mazzeh Saint, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pace R, Giuliani V, Pini Prato L, Baccetti T, Pagavino G. Apical plug technique using mineral trioxide aggregate: results from a case series. Int Endod J. 2007 Jun;40(6):478-84. doi: 10.1111/j.1365-2591.2007.01240.x. PMID 17403040
- [Result] Kandemir Demirci G, Kaval ME, Guneri P, Caliskan MK. Treatment of immature teeth with nonvital pulps in adults: a prospective comparative clinical study comparing MTA with Ca(OH)2. Int Endod J. 2020 Jan;53(1):5-18. doi: 10.1111/iej.13201. Epub 2019 Sep 3. PMID 31397907
- [Result] Alsayed Tolibah Y, Kouchaji C, Lazkani T, Abbara MT, Jbara S, Baghdadi ZD. Dental Care for a Child with Congenital Hydrocephalus: A Case Report with 12-Month Follow-Up. Int J Environ Res Public Health. 2021 Jan 29;18(3):1209. doi: 10.3390/ijerph18031209. PMID 33572890
- [Result] Vidal K, Martin G, Lozano O, Salas M, Trigueros J, Aguilar G. Apical Closure in Apexification: A Review and Case Report of Apexification Treatment of an Immature Permanent Tooth with Biodentine. J Endod. 2016 May;42(5):730-4. doi: 10.1016/j.joen.2016.02.007. Epub 2016 Mar 16. PMID 26994597
- [Result] Ajram J, Khalil I, Gergi R, Zogheib C. Management of an Immature Necrotic Permanent Molar with Apical Periodontitis Treated by Regenerative Endodontic Protocol Using Calcium Hydroxide and MM-MTA: A Case Report with Two Years Follow Up. Dent J (Basel). 2019 Jan 1;7(1):1. doi: 10.3390/dj7010001. PMID 30609673
- [Result] Khetarpal A, Chaudhary S, Talwar S, Verma M. Endodontic management of open apex using Biodentine as a novel apical matrix. Indian J Dent Res. 2014 Jul-Aug;25(4):513-6. doi: 10.4103/0970-9290.142555. PMID 25307919